CLINICAL TRIAL: NCT01115842
Title: Intervention Study Measuring Inflammatory Cytokine Levels in the Serum of Patients Who Underwent an Acute MI, and the Influence of Vitamin D on These Levels
Brief Title: Vitamin D and Inflammatory Cytokine Levels After Acute Myocardial Infraction (MI)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Arnson Yoav, MD, Clalit Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MMC10184-2009CTIL
Record Dates: First submitted 2010-05-02; First posted 2010-05-04 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-04

CONDITIONS: Acute Coronary Syndrome; Cytokines
Keywords: Vitamin D; Acute coronary syndrome; inflammatory cytokines
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): The patients will be given Vitamin D - 4000IU per day for 5 days (Day 1 through 5)
  Interventions: Drug: Vitamin D
- control (No Intervention)

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 4000IU per day for 5 days
  Arms: Vitamin D

SUMMARY:
Vitamin D is known to have immune-modulator effects including suppression of proinflammatory cytokine expression and regulation of immune cell activity. Vitamin D supplementation has been associated with a reduction in pro-inflammatory cytokines in patients with heart failure, and vitamin D deficiency has been associated with higher rates of myocardial infarcts. The levels of pro and anti-inflammatory cytokines also effect the outcome after acute coronary events.

The proposed interventional study is targeted as a feasibility study targeted at assessing the role of vitamin D as an anti-inflammatory mediator.

The study is planned as a randomized open label interventional trial. The study will be conducted of 50 adult patients (25 interventional group, 25 control), all from the internal ward in "Meir" medical center. Patients which are admitted after an acute coronary event will be randomized to the Vitamin D supplementation group or to the control group. the vitamin D group will receive 4000IU per day of vitamin D for five days. Cytokine levels will be measured at day 1 and at day 5. follow up will be continued for 6 months

Primary end point:

Levels of immune mediating cytokines (CRP, TNF-α. Il-2, IL-6, IL-12 and IL-10) after a five day intervention in patients serum.

Secondary endpoints:

Any major cardiovascular event within follow-up period. Any death of any cause during follow-up period

Expected results:

the investigators expect vitamin D supplementation after a pro-inflammatory state such as an acute coronary event, combined with conventional therapy, to result in decreased levels of inflammatory serum bio-markers.

DETAILED DESCRIPTION:
Inclusion criteria:

* Acute coronary syndrome (as defined previously).
* No advanced renal disease (creatinine levels < 1.8 for men and 1.5 for women).
* No known parathyroid or calcium homeostasis abnormalities
* Baseline Calcium levels within normal limits.
* No vitamin D supplementation taken within 4 months of current admission.
* No coexisting pro-inflammatory conditions (e.g. infection, active autoimmune disease)
* No coexisting immune-mediator agents (e.g. corticosteroids, anti-TNF or other biological agents).
* No participation in other interventional studies.
* Signing an informed consent form.

Exclusion criteria:

* Advanced renal failure
* Abnormal serum calcium levels upon admission
* Primary parathyroid or calcium homeostasis abnormalities.
* Coexisting pro-inflammatory conditions (e.g. infection, active autoimmune disease)
* Coexisting immune-mediator agents (e.g. corticosteroids, anti-TNF or other biological agents)
* Participation in other interventional studies.
* Inability or refusal to sign an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (as defined previously).
* No advanced renal disease (creatinine levels < 1.8 for men and 1.5 for women).
* No known parathyroid or calcium homeostasis abnormalities
* Baseline Calcium levels within normal limits.
* No vitamin D supplementation taken within 4 months of current admission.
* No coexisting pro-inflammatory conditions (e.g. infection, active autoimmune disease)
* No coexisting immune-mediatory agents (e.g. corticosteroids, anti-TNF or other biological agents).
* No participation in other interventional studies.
* Signing an informed consent form.

Exclusion Criteria:

* Advanced renal failure
* Abnormal serum calcium levels upon admission
* Primary parathyroid or calcium homeostasis abnormalities.
* Coexisting pro-inflammatory conditions (e.g. infection, active autoimmune disease)
* Coexisting immune-mediator agents (e.g. corticosteroids, anti-TNF or other biological agents)
* Participation in other interventional studies.
* Inability or refusal to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
inflammatory cytokine levels | 5 days of treatment
  CRP, TNF-α. Il-2, IL-6, IL-12 and IL-10

SECONDARY OUTCOMES:
MACE and all cause mortality | within 6 months
  Major acute coronary events (MACE)include:
  * revascularization
  * acute coronary syndrome
  * unstable angina pectoris

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Arnson, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel